CLINICAL TRIAL: NCT04216407
Title: The Effects Of Remote Organ Ischemic Preconditioning On Systemic Inflammatory And Glycocalyx Integrity Parameters In Living-Donor Liver Transplantation Patients
Brief Title: The Effects Of Remote Organ Ischemic Preconditioning On Systemic Inflammatory And Glycocalyx Integrity Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2019-01/02
Record Dates: First submitted 2019-12-25; First posted 2020-01-02 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Remote Organ Ischemic Preconditioning
Keywords: Remote organ ischemic preconditioning; Ischemia reperfusion injury; Glycocalyx integrity parameters; Systemic inflammation parameters
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Ischemic Preconditioning (Experimental): Short-term tourniquet on to the lower extremity before surgery
  Interventions: Procedure: Remote ischemic preconditioning
- Control (No Intervention): No intervention

INTERVENTIONS:
Procedure: Remote ischemic preconditioning — An orthopedic tourniquet was tied to the right lower extremities of the patients in RIPC arm, and tourniquet application was performed before the anhepatic phase in 3 periods of 3 minutes with an interval of 3 minutes.
  Arms: Remote Ischemic Preconditioning

SUMMARY:
Ischemia-reperfusion (IR) injury during liver transplantation is one of the major causes of mortality and morbidity associated with transplantation. Remote organ ischemic preconditioning (RIPC) is one of the most investigated practices to reduce IR injury. In this study, for the first time in the clinic, the effect of RIPC will be evaluated via both systemic inflammation parameters and also parameters showing glycocalyx integrity, on living-donor liver recipients.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed up by Acıbadem Hospital Organ Transplantation Center
* Patients accepted to participate in the study
* Older than 18 years of age
* ASA class III
* MELD score >12
* Scheduled for elective liver transplantation surgery from a living donor

Exclusion Criteria:

* Patients undergoing re-transplantation
* Under the age of 18 years
* Patients undergoing emergency surgery
* Patients with hepatorenal or hepatopulmonary syndrome
* Patients receiving mechanical ventilation support in the ICU
* Patients refusing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Tumor necrosis factor-alpha (TNF-alpha) | Postoperative early period (6 hours after intensive care unite admission)
  Evaluation of TNF-alpha level difference between groups
Intercellular adhesion molecule-1 (ICAM-1) | Postoperative early period (6 hours after intensive care unite admission)
  Evaluation of (ICAM-1) level difference between group
Hypoxia-induced factor-1 (HIF-1) | Postoperative early period (6 hours after intensive care unite admission)
  Evaluation of HIF-1 level difference between groups
Interleukin-8 (IL-8) | Postoperative early period (6 hours after intensive care unite admission)
  Evaluation of IL-8 level difference between groups
Syndecan-1 (SDC-1) | Postoperative early period (6 hours after intensive care unite admission)
  Evaluation of SDC-1 level difference between groups
soluble Vascular cell adhesion molecule-1 (sVCAM-1). | Postoperative early period (6 hours after intensive care unite admission)
  Evaluation of sVCAM-1 level difference between groups

SECONDARY OUTCOMES:
Mortality | 7 days after surgery
  Early postoperative mortality
Liver function tests | 7 days after surgery
  Evaluation of early postoperative liver function tests; AST and ALT
Length of stay in hospital and intensive care unit | 7 days after surgery
  Evaluation of the length of stay in hospital and intensive care unit
Morbidity | 7 days after surgery
  Early postoperative complications

CONTACTS AND LOCATIONS:
Locations (1):
- Acıbadem Mehmet Ali Aydinlar University Atakent Hospital, Istanbul, Atakent, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No